CLINICAL TRIAL: NCT01799681
Title: The Effects of the Hopeful Outdoor Parkinson Exercise (HOPE) Program on Improving Balance, Gait and Functional Performance in Parkinsonian Non-fallers and Single Fallers - a Randomized Controlled Trial With 12-month Follow-up
Brief Title: The Effects of the Hopeful Outdoor Parkinson Exercise (HOPE) Program on Improving Balance Performance in Parkinsonian Non-fallers and Single Fallers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Margaret Kit Yi Mak, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: approvalletter_20110823001
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: randomised controlled trial, postural balance, rehabilitation, exercise therapy, accidental falls
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXPERIMENTAL (Experimental): a 4-week indoor and 4-week outdoor balance training with stretching, strength and functional training, Balance Dance, Modified Wing Chun, Square stepping exercise, and fall-prone activities practice
  Interventions: Behavioral: an 8-week blended indoor-outdoor exercise program
- CONTROL (Active Comparator): an eight-week training on upper limb stretching and strengthening, hand agility exercise, knot tying and Chinese calligraphy
  Interventions: Behavioral: an 8-week upper limb and hand exercise program

INTERVENTIONS:
Behavioral: an 8-week blended indoor-outdoor exercise program — stretching, strength and functional training, Balance Dance, Modified Wing Chun, Square stepping exercise, and fall-prone activities practice
  Arms: EXPERIMENTAL
Behavioral: an 8-week upper limb and hand exercise program — upper limb stretching and strengthening, hand agility exercises, knot tying and Chinese calligraphy
  Arms: CONTROL

SUMMARY:
To determine whether the 8-week Hopeful Outdoor Parkinson's Exercise (HOPE) Program would be effective in improving balance performance, physical functions, gait parameter, balance confidence, health-related quality-of-life, disease-specific motor performance and fall-related outcomes in Parkinson's disease (PD) non-fallers and single fallers.

DETAILED DESCRIPTION:
Previous studies demonstrated that multi-modal balance training program was effective in improving balance performance in people with PD. However they did not include all the balance domains and outdoor fall-prone activities have been overlooked. We designed a task- and context-specific balance training program based on the framework of the Balance Evaluation Systems Test (BESTest) to target all six balance domains including biomechanical constraints, stability limits and verticality, anticipatory postural adjustments, reactive postural responses, sensori-motor integration and dynamic gait control.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PD by a neurologist (Fahn and Elton, 1987);
* aged 30 to 85 years;
* at modified Hoehn and Yahr (H&Y) stage 1.5 to 3 (Hoehn and Yahr ,1967; Goetz et al., 2004);
* able and willing to give written consent for participation in the study;
* living at home in the community;
* able to walk independently for 30 metres with or without an assistive device.

Exclusion Criteria:

* any neurological conditions other than PD;
* significant musculoskeletal or cardiopulmonary diseases;
* other disorders that may affect balance or locomotion;
* taken any structured behavioral or exercise programs in the past 3 months
* or they are receiving regular physical rehabilitation at present;
* unstable condition on anti-parkinsonian medications;
* surgical interventions for PD;
* communication or cognitive deficits with mini-mental state examination, (MMSE) <24/30 (Folstein et al., 1975);
* a history of more than two falls in the previous 12 months.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline Balance Systems Evaluation Test total and subsection scores at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention

SECONDARY OUTCOMES:
Changes from baseline comfortable gait speed at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline dual task timed-up-and-go time at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline timed-up-and-go time at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline five-times-sit-to-stand time at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline one-leg stance time at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline Activities-specific Balance Confidence Scale at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention
Changes from baseline Parkinson's disease Questionnaire (PDQ-39) at post 4-week training, post 8-week training, 6- and 12-month follow-ups | 12 months after intervention

OTHER OUTCOMES:
Changes from baseline Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) III at post 4-week training, post 8-week training, 6-and 12-month follow-ups | 12 months after intervention
Ratios of total and injurious non-fallers to fallers | 12 months after intervention
Total and Injurious fall rates | 12 months after intervention
The time to first fall and time to first injurious fall | 12 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Margaret KY Mak, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong SAR, China

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Wong-Yu IS, Mak MK. Task- and Context-Specific Balance Training Program Enhances Dynamic Balance and Functional Performance in Parkinsonian Nonfallers: A Randomized Controlled Trial With Six-Month Follow-Up. Arch Phys Med Rehabil. 2015 Dec;96(12):2103-11. doi: 10.1016/j.apmr.2015.08.409. Epub 2015 Aug 20. PMID 26299751